CLINICAL TRIAL: NCT05140109
Title: Effectiveness Randomized Controlled Trial on Eating Disorders Group Treatment: a Cognitive Dissonance, a Mindfulness and a Person-centered Based Program
Brief Title: Trial on Three Eating Disorders Group Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Lumière Lyon 2 (Other)
Responsible Party: Principal Investigator, TURGON Roxane, Principal investigator, Université Lumière Lyon 2
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A02346-33a
Record Dates: First submitted 2021-11-05; First posted 2021-12-01 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive-dissonance based program (Experimental): Group program of 8 sessions of one hour and a half.
  Interventions: Other: Arm 1: Cognitive-dissonance based program
- Mindfulness-based program (Active Comparator): Group program of 8 sessions of one hour and a half.
  Interventions: Other: Arm 2: Mindfulness-based program
- Person-centered program (Active Comparator): Group program of 8 sessions of one hour and a half.
  Interventions: Other: Arm 3: Person-centered program

INTERVENTIONS:
Other: Arm 1: Cognitive-dissonance based program — The first four sessions focus on body image and the last four sessions on eating behavior.
  Arms: Cognitive-dissonance based program
Other: Arm 2: Mindfulness-based program — The sessions focus on different contents as body image, eating behavior and emotion regulation.
  Arms: Mindfulness-based program
Other: Arm 3: Person-centered program — The sessions are not structured. Participants can bring any subject they need to talk.
  Arms: Person-centered program

SUMMARY:
This trial aims at comparing three group treatments designed for eating disorders: a Cognitive-dissonance, a Mindfulness and a Person-centered based programs. Women with eating disorders will be recruited and randomized to one of the three programs. Participants will complete a pretest, a posttest, a 3-months follow-up and a 1-year follow-up. This trial aims to compare the programs to analyze the specific dimensions upon which each program acts. The investigators therefore made hypotheses according to the programs' theory: participants in the Cognitive-dissonance based program should experience a greater decrease in eating disorders symptoms, thin-ideal internalization and body dissatisfaction and a greater improvement in quality of life than other participants. Participants in the Mindfulness-based program should show a greater improvement in negative affect and in equanimity than other participants. Participants in the Person-Centered based program should report a greater increase in congruence than other participants.

ELIGIBILITY:
Inclusion Criteria:

* eating disorders (anorexia nervosa, bulimia nervosa or binge eating disorder) or other specified feeding or eating disorder (subthreshold of anorexia, bulimia or binge eating disorder) according to Diagnostic Statistical Manual 5
* to have no regular treatment (no more than one session per month) during the 8 weeks of the program
* participants with a Body Mass Index under 17.5 could be include in the study if they had a medical monitoring in another structure

Exclusion Criteria:

* a psychotic disorder
* a bipolar disorder
* a mental retardation
* to not read or speak French fluently

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Mean change in The Eating Disorders Diagnostic Interview from pretest to 1-year follow-up | From pretest to 1-year follow-up
  The minimum of the scale is 0 and the maximum is 276. A higher score means a worse outcome.

SECONDARY OUTCOMES:
Mean change in The Hospital Anxiety and Depression Scale from pretest to 1-year follow-up | From pretest to 1-year follow-up
  The minimum of the scale is 0 and the maximum is 42. A higher score means a worse outcome.
Mean change in the subscale "Body dissatisfaction" from the scale Eating disorders inventory-2 from pretest to 1-year follow-up | From pretest to 1-year follow-up
  The minimum of the scale is 0 and the maximum is 27. A higher score means a worse outcome.
Mean change in the Sociocultural Attitudes Towards Appearance Scale from pretest to 1-year follow-up | From pretest to 1-year follow-up
  The minimum of the scale is 0 and the maximum is 150. A higher score means a worse outcome.
Mean change in the World Health Organization Quality Of Life Scale from pretest to 1-year follow-up | From pretest to 1-year follow-up
  The minimum of the scale is 0 and the maximum is 20. A higher score means a better outcome.
Mean change in the Strathclyde Inventory measuring congruence from pretest to 1-year follow-up | From pretest to 1-year follow-up
  The minimum of the scale is 0 and the maximum is 4. A higher score means a better outcome.
Mean change in the Equanimity scale from pretest to 1-year follow-up | From pretest to 1-year follow-up
  The minimum of the scale is 0 and the maximum is 7. A higher score means a better outcome.

OTHER OUTCOMES:
Presence or absence of ancillary treatment at 3-months follow-up | At 3-months follow-up and 1-year follow-up
  A YES/NO answer
Demographic data (age) at pretest | At pretest
  Current age of the participant
Demographic data (socio-professional status) at pretest | At pretest
  Current job of the participant
Demographic data (marital status) at pretest | At pretest
  Current marital status of the participnat
Demographic data (education level) at pretest | At pretest
  Educational degree of the participant
Demographic data (Body Mass Index) at pretest | At pretest
  Current height and weight of the participant
Demographic data (duration of eating disorders symptoms) at pretest | At pretest
  Number of years since the first symptoms of eating disorders
Demographic data (treatment medical history for eating disorders symptoms) at pretest | At pretest
  Names of treatment done in the past
Demographic data (traumatic medical history) at pretest | At pretest
  A YES/NO questionnaires on potential traumatic events

CONTACTS AND LOCATIONS:
Overall Officials: Roxane Turgon, Principal Investigator — Université Lumière Lyon 2
Locations (1):
- Association Endat, Paris, France

IPD SHARING:
Plan to Share IPD: No